CLINICAL TRIAL: NCT06553586
Title: Epidemiology of Road Traffic Accidents in Riyadh Region in the Last Five Years (2019-2023)
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mubarak Mohammed Saleh Alrakah, Resident of Public Health and Community Medicine, Assiut University, Egypt, Assiut University
Other Study IDs: 04-2024-200850
Record Dates: First submitted 2024-08-12; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Epidemiology; Road (Traffic) Accident [RTA] Nos; Riyadh
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data collection — Data of the proposed study will be collected from two main sites, namely they:
  1. All emergency departments of health service outlets received the concerned victims of RTAs in Riyadh Region throughout the last five years (2019-2023). The records and documents of these hospitals will be reviewed and the researcher will determine and pick up the victims of RTAs only and record them in a relevant form designed to fit with the proposed study.
  2. The General Administration of Traffic in Riyadh Region.

SUMMARY:
The findings arising from the proposed study will spot light on the issue of road traffic accidents in Riyadh Region which will help stakeholders to design proper plans and strategies of prevention and control of this issue. This will minimize the toll and burden of road traffic accidents in Riyadh Region.

To highlight the magnitude of the problem of road traffic accidents in Riyadh Region in the last five years (2019-2023), To identify the demographic characteristics of the victims involved in accidents throughout the last five years in Riyadh Region, To estimate the trend and seasonal variations of road traffic accidents Riyadh Region.

DETAILED DESCRIPTION:
Road traffic accidents (RTAs) have become a significant public health concern that requires quick attention. RTAs cause the bulk of hospital admissions due to trauma globally. The incidence of trauma caused by RTA was the highest cause of trauma-related admission (62.5%). These RTAs have the potential to cause harm to one or more bodily parts, and in extreme circumstances, they may even be fatal. They are a major contributor to early-life impairment and death. Saudi Arabia has the greatest RTA-associated mortality. RTAs account for 13% of the Saudi population's disability-adjusted life years (DALYs).

The World Health Organization (WHO) estimates that 1.25 million people die in RTAs each year, despite constant attempts to lessen the toll of these incidents on healthcare systems. Twenty to fifty million individuals experience non-fatal injuries, such as trauma and disability, necessitating extended hospital admissions. By 2030, road traffic accidents are predicted to rank the seventh cause of mortality, if the ongoing efforts to enhance healthcare are not made.

Depending on the kind of harm, RTIs can be classified into several categories. RTIs can be of any kind, ranging from cuts, piercings, and crush wounds to internal organ damage, fractures, and amputations. These injuries might impact almost any part of the body. The lower limbs were the most damaged body region in victims of RTAs, followed by the chest, upper limbs, head, and spine, as concluded by a study done between July 2014 and July 2017.

According to different researches, bigger, substantial organs, including the spleen, liver, and kidneys, are most frequently harmed by intra-abdominal lesions brought on by RTAs. There may be several pros to this classification of RTI frequency based on the type of injury and the body location impacted. According to a published research, individuals with serious brain and pelvic injuries have a high death risk. As a result, the clinicians working in the emergency room could better assess the seriousness of each individual emergency case and properly prioritize them.

ELIGIBILITY:
Inclusion Criteria:

-All the Road Traffic Accidents victims; who attended the emergency room or admitted to the hospital during the study period.

Exclusion Criteria:

-Any injury on the road without involvement of a vehicle (e.g. a person slipping and falling on the road and sustaining injury) or injury involving a stationary vehicle (e.g. persons being injured while washing or loading a vehicle).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This cross section study will be conducted on all the Road Traffic Accidents victims; who attended the emergency room or admitted to the hospital during the study period
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Road Traffic Accidents | Five years from the start of the study
  Prevalence of Road Traffic Accidents will be recorded in the Riyadh Region in the Last Five Years.

SECONDARY OUTCOMES:
Causes of Road Traffic Accidents | Five years from the start of the study
  Causes of Road Traffic Accidents will be recorded such as dangerous overtaking / lane cutting, drunken driving, over crowding and over loading, lack of driving skills and inadequate knowledge of traffic discipline.
Complication | Five years from the start of the study
  Complication will be recorded such as physical injuries, psychological trauma, financial strain, legal issues, and disruptions to traffic flow.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.